CLINICAL TRIAL: NCT00001294
Title: Genetic Factors and Interrelationships for Sexual Orientation, Susceptibility to HIV and Kaposi's Sarcoma, Alcoholism and Psychological Traits, and Histocompatibility Antigens
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920078; 92-C-0078
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-04

CONDITIONS: Alcoholism; HIV Infection; Homosexuality; Kaposi's Sarcoma
Keywords: Genetic Linkage; Sex Behavior; AIDS; Alcohol Dependence; HLA System; Cancer
MeSH Terms: conditions — Alcoholism; HIV Infections; Homosexuality; Sarcoma, Kaposi; Sexual Behavior; Acquired Immunodeficiency Syndrome; Neoplasms

SUMMARY:
We propose to test, by DNA linkage analysis of family pedigree members, the following interrelated hypotheses: 1) that sexual orientation is genetically influenced; 2) that the development of Kaposi's sarcoma and other outcomes of HIV infection in male homosexuals is affected by host susceptibility genes, circulating sex hormone levels, or HLA haplotype; and 3) that alcoholism and other psychobehavioral conditions are associated with homosexuality on a genetic basis and/or influenced by candidate behavioral loci. The subjects for these studies will be self-identified male and female homosexual probands and their relatives from families in which there are at least two individuals with homosexual orientation. All subjects will be adults, and will be referred through NIH physicians, private practitioners, and gay and lesbian organizations. Subjects will undergo a sexual orientation and behaviors interview, a psychiatric interview, and phlebotomy for HIV testing, HLA determination, endocrine measurements, and preparation of DNA from cultured lymphocytes. The DNA samples will be analyzed for a series of genetic markers that span the human genome and for candidate loci chosen for function.

DETAILED DESCRIPTION:
We propose to test, by DNA linkage analysis of family pedigree members, the following interrelated hypotheses: 1) that sexual orientation is genetically influenced; 2) that the development of Kaposi's sarcoma and other outcomes of HIV infection in male homosexuals is affected by host susceptibility genes, circulating sex hormone levels, or HLA haplotype; and 3) that alcoholism and other psychobehavioral conditions are associated with homosexuality on a genetic basis and/or influenced by candidate behavioral loci. The subjects for these studies will be self-identified male and female homosexual probands and their relatives from families in which there are at least two individuals with homosexual orientation. All subjects will be adults, and will be referred through NIH physicians, private practitioners, and gay and lesbian organizations. Subjects will undergo a sexual orientation and behaviors interview, a psychiatric interview, and phlebotomy for HIV testing, HLA determination, endocrine measurements, and preparation of DNA from cultured lymphocytes. The DNA samples will be analyzed for a series of genetic markers that span the human genome and for candidate loci chosen for function.

ELIGIBILITY:
INCLUSION CRITERIA:

The basic criterion for entering families into the DNA linkage study is the presence of two or more homosexual siblings of the same sex. Additional criteria will be imposed depending on the aims of the particular project.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 1992-01; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Pillard RC, Weinrich JD. Evidence of familial nature of male homosexuality. Arch Gen Psychiatry. 1986 Aug;43(8):808-12. doi: 10.1001/archpsyc.1986.01800080094012. PMID 3729676
- [Background] Bailey JM, Pillard RC. A genetic study of male sexual orientation. Arch Gen Psychiatry. 1991 Dec;48(12):1089-96. doi: 10.1001/archpsyc.1991.01810360053008. PMID 1845227
- [Background] Whitam FL, Diamond M, Martin J. Homosexual orientation in twins: a report on 61 pairs and three triplet sets. Arch Sex Behav. 1993 Jun;22(3):187-206. doi: 10.1007/BF01541765. PMID 8494487